CLINICAL TRIAL: NCT03892629
Title: Baduanjin Exercise for Patients With GOLD 2-3 Stable Chronic Obstructive Pulmonary Disease on Pulmonary Rehabilitation: A Prospective, Randomized, Controlled Clinical Trial
Brief Title: Baduanjin Exercise for Patients With GOLD 2-3 Stable COPD on Pulmonary Rehabilitation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: ShuGuang Hospital (Other)
Collaborators: Shanghai Zhongshan Hospital (Other)
Responsible Party: Principal Investigator, Sun Meng, Attending Physician, ShuGuang Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2018YFC1313601003
Record Dates: First submitted 2019-03-26; First posted 2019-03-27 (Actual); Last update posted 2019-04-01 (Actual); Status verified 2019-03

CONDITIONS: Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Baduanjin exercise group (Experimental): Participants in this group received Baduanjin exercise
  Interventions: Behavioral: Baduanjin exercise
- Instrument rehabilitation group (Active Comparator): Participants in this group received rehabilitation by using tri-ball respiratory trainer
  Interventions: Device: Instrument rehabilitation
- Baduanjin Exercise and Instrument Rehabilitation (Active Comparator): Participants in this group received both instrument rehabilitation and Baduanjin exercise
  Interventions: Behavioral: Baduanjin exercise; Device: Instrument rehabilitation
- No Intervention (No Intervention): Participants in this group only received routine drug-treatment

INTERVENTIONS:
Behavioral: Baduanjin exercise — Participants received Baduanjin exercise. Each Baduanjin exercise session lasts 30 minutes and continues twice a day, 5 times per week for 12 weeks
  Arms: Baduanjin Exercise and Instrument Rehabilitation; Baduanjin exercise group
Device: Instrument rehabilitation — Participants received pulmanory rehabilitation by using tri-ball respiratory trainer. Each instrument exercise session lasts 30 minutes and continues twice a day, 5 times per week for 12 weeks
  Arms: Baduanjin Exercise and Instrument Rehabilitation; Instrument rehabilitation group

SUMMARY:
Chronic Obstructive Pulmonary Disease (COPD) is a disease with a very high morbidity and mortality rate. When the lung function drops lower and lower, patients will bear great affliction physically and mentally. How to improve the quality of life in patients with COPD is a hot topic in the study of COPD now. Baduanjin, as one of the traditional Chinese qigong exercises, has the features of generous stretch, soft consistency, dynamic but static, which is an appropriate movement pattern for COPD patients.

DETAILED DESCRIPTION:
To investigate the efficacy of Baduanjin exercise for patients with stable chronic obstructive pulmonary disease on phase II~III. A prospective, randomized, controlled clinical trial was designed.

ELIGIBILITY:
Inclusion Criteria:

* Aged from 40 to 80 years
* Diagnosed with stable chronic obstructive pulmonary disease
* Phase II~III

Exclusion Criteria:

* The condition was serious or movement restrained by other diseases
* In the acute exacerbation of chronic obstructive pulmonary disease
* Participants who have contraindications to exercise training
* Patients who have other serious acute, chronic organic disease or mental disorders

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2019-04 (Estimated); Primary Completion 2019-10 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
St. George's respiratory questionnaire (SGRQ) | Baseline, 3 months, 6 months
  Evaluating the changes of impact on quality of life
Six-minute walk test (6MWT) | Baseline, 3 months, 6 months
  Testing patients changes on walking distance and accompanies symptoms in 6 minutes

SECONDARY OUTCOMES:
Pulmanory function indicators (FEV1/FVC, FEV1pred%) | Baseline, 3 months, 6 months
  Assessing changes of airway limitation
Modified British medical research council questionnaire (mMRC) | Baseline, 1 month, 2 months, 3 months, 6 months
  Evaluating the severity of dyspnea, totally has 5 grade from 0-4, the higher grade represent a severer symptom
COPD assessment test (CAT) | Baseline, 1 month, 2 months, 3 months, 6 months
  Assessing the quality of life, the total score ranges from 0-40, the higher score represent a worse outcome
Times of acute exacerbation | Baseline, 1 month, 2 months, 3 months, 6 months
  Recording the frequency of acute exacerbation
Self-rating anxiety scale (SAS) | Baseline, 3 months, 6 months
  Evaluating the stage of anxiety, the total score ranges from 20-80, the higher score represent a worse outcome
Self-rating depression scale (SDS) | Baseline, 3 months, 6 months
  Evaluating the stage of depression, the total score ranges from 20-80, the higher score represent a worse outcome

OTHER OUTCOMES:
The main TCM symptoms | Baseline, 1 month, 2 months, 3 months, 6 months
  The changes of scores of TCM syndromes, the total score ranges from 0-15, the higher score represent a worse outcome

CONTACTS AND LOCATIONS:
Overall Officials: Wei Zhang, Master, Study Chair — Shanghai Shuguang Hospital
Locations (1):
- Shanghai Shuguang Hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: No